CLINICAL TRIAL: NCT04015258
Title: Metabolic Mechanisms Underlying the Responsiveness to Blueberry Interventions Aimed at Improving Cognition and Peripheral Blood Flow
Brief Title: Blueberry Study Aimed at Improving Cognition and Peripheral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Research Ethics 10113
Record Dates: First submitted 2019-03-04; First posted 2019-07-10 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-07

CONDITIONS: Vascular Stiffness; Cognitive Change; Blood Pressure
Keywords: blueberry; intervention; endothelial function; cognition; metabolomics; genomics
MeSH Terms: interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blueberries (Experimental): Fresh blueberries purchased from local supermarket will be distributed to each participant for 1 week's consumption, 160 grams per day
  Interventions: Dietary Supplement: Blueberries
- Blueberry powder (Experimental): Freeze-dried blueberry powder will be distributed to each participant for 1 week's consumption, 20 grams per day, equivalent to 160 grams of fresh blueberries
  Interventions: Dietary Supplement: Blueberry powder
- Blueberry components capsules (Placebo Comparator): Encapsulated microcrystalline cellulose powder will be blinded as blueberry components capsules to be distributed to each participant for 1 week's consumption
  Interventions: Dietary Supplement: Blueberry components capsules

INTERVENTIONS:
Dietary Supplement: Blueberries — fresh spanish blueberries
  Arms: Blueberries
Dietary Supplement: Blueberry powder — freeze-dried blueberry powder
  Arms: Blueberry powder
Dietary Supplement: Blueberry components capsules — encapsulated blueberry components (microcrystalline cellulose powder in actual)
  Arms: Blueberry components capsules

SUMMARY:
Blueberries are rich in the content of a variety of biologically active chemicals that contribute to their health properties. The consumption of blueberries has beneficial effects on vascular function and brain health and function. Blueberries are present in human diet in a number of forms, but the investigator do not know which form is best for health and why people respond differently to eating blueberries.

The aim of the present study is to assess the effects of 1 week's supplementation of whole blueberries or freeze-dried blueberry powder or encapsulated blueberry components on vascular function and brain health and function. Investigators will then categorise participants as those who have large effects of the intervention (responders) and those that don't show much effect at all (non-responders). Then the investigators will look into the role that genes play in this response and determine if metabolism is similar in these groups of participants. Any changes in participants' brain health and vascular function will be linked to these metabolic and genomic pathways, and this will help the investigators to further understand how blueberry consumption can benefit human health.

DETAILED DESCRIPTION:
Study design: The present study will supply either 160 g of fresh whole blueberry (4 handful portion) or 20 g of freeze-dried blueberry powder (measured with tablespoon provided; equivalent to 160 g of whole fresh blueberry), or placebo capsule with only microcrystalline cellulose (approx. 10 g, they will be blinded that this is encapsulated blueberry extract components) to 80 subjects on separate occasions with age range of 18-60 years old for 1 week with 1 week of washout period. Fresh blueberries will be purchased from local supermarkets; freeze-dried blueberry powder will be purchased from Lio-Licious freeze-dried fruits range; the microcrystalline cellulose will be purchased from Blackburn Distributions. There is no outside interest that could constitute commercial conflict of interest.

Methodology and sampling strategy: a randomised crossover design will be implemented. The study is a quantitative experiment and participants will be recruited through opportunity sampling.

Data collection: On each visit, cognition data will be obtained from computerised testing system COMPASS. Blood pressure will be obtained using fully automatic oscillometric device. On visits 2-7, PWV value is obtained by SphygmoCor; untargeted metabolomics and genomic data will be obtained from blood and urine sample collection.

For data analysis: The identification of responders to the treatments will be done by the calculation of response level first: response level = (change from baseline score/baseline score) x 100%. The calculated percentage will be used to characterise subjects from lowest response to highest response level. The association among -omics biomarkers and cognitive tests/endothelial parameters, lipid status under each treatment will be analysed using linear regression models after adjusting for confounding factors like age. Pathway analysis will be used to identify metabolic pathways that characterise responders and non-responders. Pathways will be identified using discriminatory metabolites from metabolomics and SNP analysis.

ELIGIBILITY:
Inclusion Criteria:

* Interested in taking part in the study
* Healthy
* Aged 18-60 years (inclusive)

Exclusion Criteria:

* Smoking
* Aged under 18 or over 60
* Blood Pressure ≥ 145/100 mmHg and are taking medication
* Have vascular disease, or other cardiac abnormalities
* Have previously suffered any head injuries, history of seizures or other neurological disorders
* Have any metabolic disorders, malabsorption syndromes or gastrointestinal complications
* Current use of above disease relevant prescription medications (excluding contraception)
* Irregular bowel function (less than 1 bowel movement per day)
* Regularly consume blueberries/blueberry-contained products more than twice per week
* Have regularly used nutritional supplements or medications within the previous 3 months (defined as more than 3 consecutive days or 4 days in total)
* Learning difficulties and dyslexia
* Visual impairment that cannot be corrected with glasses or contact lenses including colour blindness
* Currently suffer from migraines (> 1 per month)
* Body mass index (BMI) under 18.5 or over 30
* Pregnancy, seeking to become pregnant, or current lactation
* Inability to complete all of the study assessments
* Current participation in other clinical or nutrition intervention studies
* Not proficient in English equivalent to IELTS band 6 or above
* Have any known active infections

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of participant recalling word list Immediately | 1 minute
  will be assessed via COMPASS (Computerised Mental Performance Assessment System) tasks by participants recalling word list immediately after displays; the result will be presented as accuracy (%) and as an assessment of short-term memory
Correct responses of participants counting down from certain number by subtracting 3 | 5 minutes
  will be assessed via COMPASS tasks by participants counting down from certain number by threes. The result will be presented as correct responses and as an assessment of executive function
Correct responses of participants counting down from certain number by subtracting 7 | 5 minutes
  will be assessed via COMPASS tasks by participants counting down from certain number by sevens, the result will be presented as correct responses and as an assessment of executive function
Reaction time of participants' vigilance during rapid visual tracking and accurate selection of target digit stimuli | 5 minutes
  will be assessed via COMPASS tasks by measuring participants' vigilance during rapid visual tracking and accurate selection of target stimuli, presented by reaction time in millisecond (ms), as an assessment of attention and psychomotor speed
Accuracy of participant recalling word list 30 minutes after displays | 5 minutes
  will be assessed via COMPASS tasks by participants recalling word list after 30 minutes, the result will be presented as accuracy (%) and as an assessment of memory
Brachial-radial distance | 1 minute
  brachial-radial distance in meters (m), will be measured by tape
Pulse wave time | 10 minutes
  time of the pulse wave moves down from brachial to radial artery in seconds (s), will be measured by Sphygmocor (ScanMed medical)
Pulse wave velocity (PWV) | 10 minutes
  will be measured by Sphygmocor (ScanMed medical), by outcome 7 pulse wave time (s) dividing outcome 6 brachial-radial distance (m), PWV will be presented in the units of m/s, as an assessment of endothelial function
Blood Pressure | 10 minutes
  will be assessed by BP monitor and reported in the units of mm Hg

SECONDARY OUTCOMES:
Inter-cellular Adhesion Molecules (ICAMs) and Vascular Cell Adhesion Molecules (VCAMs) | 1 day
  Endothelial dysfunction's biomarkers (ICAMs and VCAMs) assessed by ELISA Kits and reported in the units of U/mL
C-reactive Protein (CRP) | 1 day
  Endothelial dysfunction's biomarkers (CRP) assessed by ELISA Kits in the units of mg/L
Plasma Lipid Status | 1 day
  Total and High-density lipoprotein (HDL-), Low-density lipoprotein (LDL-) cholesterol and triglycerides assessed by outsourcing to the local hospital, the results will be reported in the units of mmol/L
Untargeted Plasma and Urine Metabolites | 1 day
  liquid-chromatography mass spectrometry-based techniques (LCMS) will be applied to identify untargeted metabolites in the plasma and urine samples
Single Nucleotide Polymorphisms (SNPs) | 7 days
  SNP arrays will be applied for genotyping participants' DNA collected from the buffy coat of the blood sample, following the removal of plasma

CONTACTS AND LOCATIONS:
Overall Officials: Yueyue Wang, Principal Investigator — Miss
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No